CLINICAL TRIAL: NCT05164055
Title: A French Multicenter Open Label Phase 4 Extension Study of Long-term Safety and Efficacy in Patients With Pompe Disease Who Previously Participated in Avalglucosidase Alfa Development Studies in France
Brief Title: Avalglucosidase Alfa French Post-trial Access for Participants With Pompe Disease (PTA Avalglucosidase)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTA17333; U1111-1266-5434 (Registry Identifier: ICTRP); 2024-514773-22 (Registry Identifier: CTIS); 2021-002590-26 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-12-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avalglucosidase alfa (Experimental): Administered intravenously every other week
  Interventions: Drug: Avalglucosidase alfa (GZ402666)

INTERVENTIONS:
Drug: Avalglucosidase alfa (GZ402666) — Pharmaceutical form: Sterile lyophilized powder Route of administration: intravenous (IV) infusion
  Other Names: Nexviadyme®

SUMMARY:
This long-term open label safety and efficacy study is intended to follow up, and to provide post-trial access to enzyme replacement therapy (ERT) with avalglucosidase alfa to patients with Pompe disease in France who have completed Study EFC14028, LTS13769, or ACT14132, from market authorization until reimbursement of avalglucosidase alfa in France or until September 2026, whichever comes first.

- Study visit frequency: every 2 weeks

DETAILED DESCRIPTION:
Treatment duration approximately 4 years and 3 months: until reimbursement of avalglucosidase alfa in France or until September 2026, whichever comes first

ELIGIBILITY:
Inclusion Criteria:

* Patient with LOPD or IOPD who has previously completed Study EFC14028, LTS13769, or ACT14132 in France, and reimbursement for avalglucosidase alfa is not yet granted in France.
* The patient and/or their parent/legal guardian is willing and able to provide signed informed consent, and the patient, if <18 years of age, is willing to provide assent if deemed able to do so.
* The patient (and patient's legal guardian if patient is <18 years of age) must have the ability to comply with the clinical protocol.
* The patient, if female and of childbearing potential, must have a negative pregnancy test result [urine beta-human chorionic gonadotropin (β-HCG)] at enrollment.
* Sexually active female patients of childbearing potential and male patients are required to practice true abstinence in line with their preferred and usual lifestyle or to use 2 acceptable effective methods of contraception.

Exclusion Criteria:

* Patient with life-threatening hypersensitivity (anaphylactic reaction) to one of avalglucosidase alfa's excipients.
* Patient who permanently discontinued avalglucosidase alfa in a previous clinical study
* Pregnant or breastfeeding female patient
* The patient is concurrently participating in another clinical study of investigational treatment.
* The patient, in opinion of the Investigator, is unable to comply with the requirements of the study.
* The patient has clinically significant organic disease (with the exception of symptoms relating to Pompe disease), including clinically significant cardiovascular, hepatobiliary, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precludes participation in the study or potentially decreases survival.
* Individuals accommodated in an institution because of regulatory or legal order; prisoners, or patients who are legally institutionalized.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE), treatment-emergent adverse events (TEAE), including infusion associated reactions (IAR) and death | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months

SECONDARY OUTCOMES:
Assessment of six-minute walk test (distance in meters and % predicted value) for late-onset Pompe disease (LOPD) and infantile-onset Pompe disease (IOPD) participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  The primary measurement is the distance in meters walked by the participant on a flat, hard surface in 6 minutes. The distance walked in meters will be recorded and the corresponding percent predicted value will be calculated. The greater the distance (that a participant could walk in 6 minutes), the greater the endurance.
Assessment of quick motor function test (QMFT) for LOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  The QMFT is an observer administered test to evaluate changes in motor function. QMFT comprises of 16 items specifically difficult for participants with Pompe disease. Each item is scored separately on a 5-point ordinal scale (ranged from 0 to 4, higher score indicated better outcome). Total QMFT score is obtained by adding the scores of all items and ranged from 0 (unable to perform motor function tests) to 64 (normal muscle function), higher score represented better outcome.
Pulmonary function tests (forced vital capacity [FVC] (% predicted), maximum expiratory pressure/maximum inspiratory pressure) in upright and supine positions for LOPD and IOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position, also tested in supine position. Percent of predicted FVC = (actual FVC measurement)/(predicted value of FVC) * 100.
  Maximum Inspiratory Pressure (MIP) is a quick and non-invasive test to measure strength of inspiratory muscles, primarily diaphragm, and allows for assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MIP refers to how much air pressure force an individual creates by inhaling through the mouth as hard as possible.
  Maximum Expiratory Pressure (MEP) is a quick and non-invasive test to measure strength of expiratory muscles, primarily diaphragm, and allows for assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MEP is the greater pressure generated during maximal expiration.
Quality of life evaluation: 12-item short form health survey (SF-12) for LOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  SF-12, a 12 item-questionnaire, used to assess health-related quality of life in participants aged >=18 years at screening/baseline. SF-12 consisted of 12 items, which were categorized into eight domains (subscales) of functioning and well-being: physical functioning, role-physical, role emotional, mental health, bodily pain, general health, vitality and social functioning, with each domain score ranged from 0 (poor health) to 100 (better health), higher scores indicated good health condition. These eight domains were further summarized into 2 summary scores, physical component summary (PCS) and mental component summary (MCS). The score range for each of these 2 summary scores was from 0 (poor health) to 100 (better health), higher scores indicated a better health-related quality of life.
Quality of life evaluation: Pompe Disease Symptom Scale (PDSS) for LOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  The 24-hour recall PDSS (V1.1) is a self-administered questionnaires specifically designed to capture the symptoms impacts relevant to patients with LOPD. The PDSS includes 12 questions with responses on a scale from 0 (none) to 10 (as bad as I can imagine) The data from PDSS scale will be analyzed separately and as a composite with PDIS scale.
Quality of life evaluation: Pompe Disease Impact Scale (PDIS) for LOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  The 24-hour recall PDIS (V1.2) is a self-administered questionnaires specifically designed to capture disease impacts relevant to patients with LOPD. The PDIS includes 15 questions with varying scales implemented depending on question type. The data from PDIS scale will be analyzed separately and as a composite with PDSS scale.
Pompe Pediatric Evaluation of Disability Inventory (Pompe-PEDI) score for IOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  The Pompe-PEDI consists of a Functional Skills Scale and a Caregiver Assistance Scale. Both scales have 3 domains: self-care; mobility; and social function. The Mobility Domain was selected to measure change in mobility secondary to changes in muscle strength. The domain consists of 160 mobility items.
PedsQL score for IOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  The 23item PedsQL Generic Core Scale encompasses 4 subscales including physical, emotional, school, and social functionings. Scores are transformed to a 0-100 scale, higher scores indicate better HRQOL.
  Infant scale will not be used since this is a scale for up to 24 months of age and patients are older now than that.
Left Ventricular Mass Index (LVMI) Z-score in IOPD participants | From study enrolment to the final study visit/telephone contact, up to 4 years and 3 months (at enrolment and every 6 months)
  Left Ventricular Mass Index (LVMI) equivalent to mean age specific LVMI plus 2 standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- France (11):
  - Investigational Site Number : 2500004, Bordeaux
  - Investigational Site Number : 2500005, Brest
  - Investigational Site Number : 2500008, Clermont-Ferrand
  - Investigational Site Number : 2500009, Lille
  - Investigational Site Number : 2500003, Lyon
  - Investigational Site Number : 2500001, Marseille
  - Investigational Site Number : 2500006, Nantes
  - Investigational Site Number : 2500007, Nice
  - Investigational Site Number : 2500002, Paris
  - Investigational Site Number : 2500010, Paris
  - Investigational Site Number : 2500011, Tours

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PTA17333 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25338&tenant=MT_SNY_9011